CLINICAL TRIAL: NCT01615328
Title: Evaluation of Fusion Rate of Anterior Cervical Discectomy and Fusion (ACDF) Using Cervios ChronOs™ and Bonion™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bonion ACDF
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Intervertebral Disk Degeneration; Intervertebral Disk Displacement; Ossification of Posterior Longitudinal Ligament
Keywords: anterior cervical discectomy and fusion; bone graft substitute; PEEK cage; hydroxyapatite; demineralized bone matrix; b-tricalcium phosphate; Bonion; Cervios ChronOs
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Ossification of Posterior Longitudinal Ligament

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervios ChronOs (Experimental): The ACDF surgery will be carried out with Cervios ChronOs(TM), which is the PEEK cage filled with b-TCP.
  Interventions: Device: Cervios ChronOs
- Bonion (Experimental): The ACDF surgery will be carried out with Bonion(TM), which is the PEEK cage with HA/DBM.
  Interventions: Device: Bonion

INTERVENTIONS:
Device: Cervios ChronOs — The ACDF surgery will be carried out with Cervios ChronOs after randomization procedure.
  Arms: Cervios ChronOs
Device: Bonion — The ACDF surgery will be carried out with Bonion after randomization procedure.
  Arms: Bonion

SUMMARY:
Anterior cervical discectomy and fusion (ACDF) has shown good treatment results for a variety of cervical spine diseases such as herniated intervertebral disc (HIVD), cervical spondylotic radiculopathy (CSR) and cervical spondylotic myelopathy (CSM). ACDF using autogenous iliac bone graft is gold standard, however, it may lead to donor-site morbidities. Preventing these complications, some authors have tried to use alterative bone graft substitutes. Among these alternatives, Cervios ChronOs™ which is the polyetheretherketone (PEEK) cage with b-tricalcium phosphate (TCP) has become popular and shown good clinical results. However, b-TCP has only osteoconduction ability of three osteogenic properties.

Recently, Bonion™ which is the PEEK cage filled with hydroxyapatite (HA) / demineralized bone matrix (DBM) is introduced. HA/DBM mixture has abilities of osteoconduction and osteoinduction, therefore this alternative is expected to show superior bone fusion capability to PEEK cage with b-TCP. However, there has been no comparison study between the PEEK cage with b-TCP and the PEEK cage with HA/DBM. The purpose of this study is to evaluate bone fusion rate between these cervical spine cages using postoperative computed tomography (CT)

DETAILED DESCRIPTION:
Biologically, graft material should be endowed with several basic properties. Several synthetic materials and graft substitutes have been developed to maximize fusion outcomes while avoiding complications of harvesting autograft. Mixture of hydroxyapatite (HA) and β-tricalcium phosphate (β-TCP), have been widely utilized for bony regeneration. On the other hand, demineralized bone matrix (DBM) has been utilized as a graft substitute with mainly its osteoinductive ability. While HA and β-TCP have osteoinductive osteoconductive properties and DBM has osteoconductive osteoinductive properties, a graft material fully incorporating both properties has not been developed. We hypothesize that an interbody graft material equipped simultaneously with osteoinductivity and osteoconductivity would enhance fusion achievement; however, clinical trials with mixture materials within a PEEK cage in ACDF surgery have rarely been performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervical HIVD, CSR, CSM or OPLL
* The patient who is expected to receive anterior cervical discectomy and fusion operation.
* Volunteer for this study with written consent.

Exclusion Criteria:

* Patient with cervical spine fracture, infection.
* Below -3.5 T-score by DEXA bone densitometry
* Patient with hemorrhagic diseases
* Patient with malignancy
* Patient who is not suitable for this study judged by principal investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Sup Yeom, MD, PhD, Principal Investigator — Seoul National Univerity Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervios ChronOS: The patients underwent ACDF using Cervios ChronOS(TM) which is the PEEK cage filled with b-TCP.
- Bonion: The patients underwent ACDF using Bonion which is the PEEK cage with Hydroxyapatite and demineralized bone matrix.
Period: Overall Study
Arm/Group | Cervios ChronOS | Bonion
Started | 42 | 43
Completed | 39 | 38
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervios ChronOS | Bonion | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.4) | 51.9 (11.7) | 51.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 26 | 25 | 51
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Bone Fusion With CT(Postoperative 6 Months)
Description: Evaluation of bone fusion between bone substitutes and cervical vertebral endplates with 3-dimensional CT at 6 months after operation (ACDF).
Time Frame: 6 months after surgery(ACDF)
Measure: Number; unit: participants
Arm/Group | Cervios ChronOS | Bonion
Number analyzed (Participants) | 39 | 38
participants | 26 | 28

2. Secondary Outcome: VAS of Radiating Pain (Postoperative 6 Months)
Description: Evaluation of radiating pain using the visual analogue scale (VAS) at 6 months after operation (ACDF).
  Reported pain using VAS was recorded and evaluated. Patients were instructed to make a mark on a horizontally-oriented, 10-point VAS labeled "no pain (zero point)" at the far left and "greatest pain (ten point)" at the far right.
Time Frame: at 6 months after surgery (ACDF)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cervios ChronOs | Bonion
Number analyzed (Participants) | 39 | 38
scores on a scale | 2.4 (2.3) | 2.9 (2.5)

3. Secondary Outcome: VAS of Neck Pain(Postoperative 6 Months)
Description: Evaluation of neck pain using the visual analogue scale (VAS) at 6 months after operation (ACDF).
  Reported pain using VAS was recorded and evaluated. Patients were instructed to make a mark on a horizontally-oriented, 10-point VAS labeled "no pain (zero point)" at the far left and "greatest pain (ten point)" at the far right.
Time Frame: at 6 months after surgery (ACDF)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Cervios ChronOs: The ACDF surgery will be carried out with Cervios ChronOs(TM), which is the PEEK cage filled with b-TCP.
  Cervios ChronOs: The ACDF surgery will be caried out with Cervios ChronOs after randomization procedure.
- Bonion: The ACDF surgery will be carried out with Bonion(TM), which is the PEEK cage with HA/DBM.
  Bonion: The ACDF surgery will be caried out with Bonion after randomization procedure.
Arm/Group | Cervios ChronOs | Bonion
Number analyzed (Participants) | 39 | 38
scores on a scale | 2.3 (2.4) | 2.0 (2.4)

ADVERSE EVENTS:
Arm/Group | Cervios ChronOS | Bonion
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38

LIMITATIONS AND CAVEATS:
Our study was included relatively small samples and short follow-up periods with 77 patients and one year duration. the measurement bias could be presented by individually different extent of neck flexion and extension in dynamic radiographs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less